CLINICAL TRIAL: NCT04456335
Title: Investigation of Supragingival Plaque Microbiome Using Next Generation Sequencing in Early Childhood Caries
Brief Title: Investigation of Supragingival Plaque Microbiome in Early Childhood Caries
Status: Completed | Type: Observational
Sponsor: Trakya University (Other)
Responsible Party: Principal Investigator, ŞİRİN GÜNER ONUR, Assist. Prof. Dr., Trakya University
Other Study IDs: 2018/269
Record Dates: First submitted 2020-06-18; First posted 2020-07-02 (Actual); Last update posted 2020-07-02 (Actual); Status verified 2020-06

CONDITIONS: Early Childhood Caries
Keywords: Early childhood caries; Oral Microbiome; Next generation sequencing

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Supragingival plaque sample
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Caries-free: Caries-free children
  Interventions: Genetic: Collection of supragingival plaque from caries free children
- Early childhood caries: Children with early childhood caries
  Interventions: Genetic: Collection of supragingival plaque from caries free children

INTERVENTIONS:
Genetic: Collection of supragingival plaque from caries free children — Supragingival plaque samples were collected from posterior molar teeth
  Other Names: Collection of supragingival plaque from children with early childhood caries

SUMMARY:
The purpose of this study was to characterize the supragingival plaque microbiome in children with early childhood caries and identify potential microorganisms associated with caries.

DETAILED DESCRIPTION:
Sixty children with and without early childhood caries were recruited from Trakya University Faculty of Dentistry Department of Pediatric Dentistry. Oral examinations were performed by the same examiner according to diagnostic criteria of World Health Organisation (WHO) and The International Caries Detection and Assessment System (ICDAS) . Mothers' completed a structured questionnaire on the socio-demographic informations, child's feeding practices and oral hygiene habits. After the oral examination, supragingival plaque samples were collected from the posterior tooth surfaces. Supragingival plaque samples were examined with the Illumina MiSeq new generation sequencing method.

ELIGIBILITY:
Inclusion Criteria:

* 36-71 months old children
* No history of any medical problem
* No history of antibiotic in the three months prior to sampling
* Any sign of early childhood caries,
* Caries free children
* Mothers accepted to complete a structured questionnaire
* Children who cooperate for dental examination and sample collection

Exclusion Criteria:

* Children older than 71 months
* Medically compromised
* Children with antibiotic use history at last three months
* Children refused dental examination and plaque collection
* Mothers' refused to complete questionnare

Ages: 36 Months to 71 Months | Sex: All
Age Groups: Child
Study Population: A total of sixty children with early childhood caries(n=30) and caries free(n=30)
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2019-03-04 (Actual); Primary Completion 2020-01-03 (Actual); Study Completion 2020-05-23 (Actual)

PRIMARY OUTCOMES:
V4-16S rRNA and ITS1 rRNA sequencing | 6 months
  Supragingival plaque samples were collected from the tooth surfaces using a sterile periodontal curette. DNA extraction was performed at Sugenomik Biotechnology Laboratory for library preparation and paired-end Illumina MiSeq PE250 sequencing of the V4 region of bacterial 16S rRNA and fungal ITS1 (internal transcribed spacer 1) rRNA genes.

CONTACTS AND LOCATIONS:
Locations (1):
- Trakya Universitiy Faculty of Dentistry Department of Pediatric Dentistry, Edirne, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No